CLINICAL TRIAL: NCT01383187
Title: An Open-label, Non Randomized, Single-Center Registry Study to Assess the Safety and Effects of Autologous Platelets Concentrate and Autologous Thrombin for the Treatment of Deep Burns Trauma
Brief Title: Autologous Platelets Concentrate and Autologous Thrombin for the Treatment of Deep Burn Trauma
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 99-OVZ-09-024
Record Dates: First submitted 2011-06-21; First posted 2011-06-28 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2013-03

CONDITIONS: Burns
Keywords: Deep Burn Trauma; Dermo-Epidermal Graft; Platelet Rich Plasma Concentrate (PRP); Vancouver Scar Score; Scarring; Hypertrophic Scarring
MeSH Terms: conditions — Burns; Cicatrix; Cicatrix, Hypertrophic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DE graft and PRP concentrate (Experimental): Patients enrolled in this arm receive the innovative treatment methods consisting of application of DE graft together with PRP concentrate.
  Interventions: Procedure: DE graft and PRP concentrate
- Standard treatment group (Active Comparator): PAtients included into this arm will receive a standard treatment for deep-burn injuries, i.e. DE graft without the application of the PRP concentrate.
  Interventions: Procedure: DE graft

INTERVENTIONS:
Procedure: DE graft and PRP concentrate — Application of DE graft together with PRP concentrate
  Arms: DE graft and PRP concentrate
Procedure: DE graft — DE grafting presents a standard treatment method in patients with deep-burn trauma.
  Arms: Standard treatment group

SUMMARY:
Deep skin burn injuries, especially extensive deep burns or/and deep burns extending on the face, hands, feet, genitalia and perineum, remain one of the most challenging therapeutic problems. Surgical excision of the necrotic burned tissue with subsequent skin grafting of the affected area has become the golden standard for the treatment of deep partial thickness and full thickness skin burns and represents the treatment of choice. Despite of all the progress achieved in the treatment process (artificial skin, cultured keratinocytes), the therapeutic results are sometimes unacceptable due to functional and cosmetic deficits causing severe psychological and emotional distress, particularly in the form of disfiguring and disabling scarring - i.e. hypertrophic scars, joint contractures restricted movement, peripheral neuropathy, psychiatric and physiological diseases, as well as thermoregulation disorders. Consequently, the quality of life is markedly decreased. That is why new methods of burn wounds covering are intensively searched. Based upon the results of available pre-clinical studies, the local use of autologous platelet concentrate with their active growth factors appears to be a good and promising possibility how to improve faster and higher quality of healing deep skin burn wounds.

DETAILED DESCRIPTION:
Deep skin burn injuries(i.e. third-degree and deep second-degree burns), especially extensive deep burns or /and deep burns extend on the face, hand, feet, genitalia and perineum remain one the most challenging problem for modern medicine because of its difficult, complicated and long clinical course and recovery. Extensive deep burn injury is, in despite of all progress in treatment, ordinarily associated with shock, infection, MODS, electrolyte imbalance, respiratory distress,… with high morbidity and mortality rate. Regardless of the extent,burns are likewise very painful with necessity to treat pain in the majority of patient, comprehensive treatment and wound management of deep burns often demand confinement to bed, splinting, special positioning - patients are some point of time unable care of themselves and restrict in their habitual life pattern. Despite of all the progress achieved in the treatment process, therapeutic results sometimes are unacceptable due to functional and cosmetic deficits causing severe psychological and emotional distress, particularly due to scarring and physical deformity - i.e. hypertrophic scars, joint contractures, peripheral neuropathy, psychiatric and psychological diseases, as well as thermoregulation disorders. Consequently the quality of life may be markedly decreased. That is why the new methods of burn wounds covering are intensively searched. Based upon the results of available pre-clinical studies, the local use of autologous platelet concentrate with their active growth factors appears to be a good possibility how to improve faster and higher quality of healing deep skin burn wounds.

To achieve the best possible therapeutic results the accurate diagnosis of depth of skin destruction and depending on that the accurate choice of treatment strategy is fundamental. The standard method for the determination of burn depth is clinical examination. Presence of the eschar, i.e. evidently devitalised tissue, means necessity of surgical treatment and the clinical diagnosis is obvious. The accurate clinical assessment of the deep dermal burns,which may sometimes healing spontaneously until 21 days without surgical treatment, is in most of cases complicated and controversial. If the healing until 21 days is not complete or the possibility of spontaneous healing is improbable, the surgical treatment is indicated. In these controversial cases the dominant role plays above all clinical experiences and diagnostic capabilities of examining burn´s surgeon. Indication of surgical treatment here directly depends on human factor and is related with the risk of incorrect decision. Despite of the fact that there is no generally accepted physical diagnostic method to detect the depth of burns, there are some objective methods how to improve the accuracy of diagnosis and their using in parallel with clinical observations is desirable. In our Burn centre the investigators use the laser Doppler method to determine the depth of burns by means of apparatus LDPI PIM III (Perimed Co, Jarfalla,Sweden). This device detects skin perfusion and its changes in the course of time. Third degree burns have a very low levels of skin perfusion and in course of time there is no increase of perfusion units on measured areas. Deep second degree burns with presumption of spontaneous healing within 14 - 21 days show continued increase of perfusion units from the second to ninth day post-injury. Deep second degree burns with healing time longer than 21 days show minimal or no increase of perfusion units from second to eleventh post-injury day. Current treatment of deep burns consists of surgical excision of necrotic tissue followed by dermoepidermal skin autografting. Central role of platelets in haemostatic and thrombotic process is well known. This is due to many clotting and growth factors stored in platelet granules. The successful use of the autologous platelet rich plasma (PRP), i.e. Autologous Platelet Concentrate (APC) to improve healing has been recently tested in limited in vivo and lately in a few clinical trial as well, however no published study to our knowledge has tested APC for the treatment of deep skin burns in humans. Based on data from published literature and our limited clinical experience with the use of APC to treat severe skin ulcerations, the investigators would like to use this knew experimental treatment in our patient population suffering from deep skin burns.

1. third-degree burns, i.e. full thickness burns involve all the layers of skin.
2. fourth-degree burns - when muscle, bone and blood vessels also be injured.

2/ deep second-degree burns, i.e. burns involved damage of the epidermis and deep part of the dermis layer of skin. Deep second-degree burns can sometimes heal spontaneously, however in cases when the investigators supposed the healing takes longer than three weeks, the investigators indicate surgical treatment for optimal functional and cosmetic results.

Surgical excision of devitalised burned tissue with subsequent skin grafting on the basis of longtime clinical experiences has become the golder standard for the treatment of deep partial thickness and full thickness skin burns in generally and represents the treatment of choice in our Burn center.In order to achieve the best therapeutic results,i.e. un-complicated,quick and high quality healing, the new methods of burn wounds covering are intensively searched. One of many possibilities is topical transplantation of APC, successfully used in many surgical fields about twenty years, but still widely uncertified in clinical practice of burn´s medicine.

A concentrate of autologous thrombocytes - Autologous Platelet Concentrate (APC) is applied locally in the area of autotransplanted surfaces. The applied growth factors initiate chemotaxis, proliferation, angiogenesis, proteosynthesis, reparation and remodeling of the impaired tissue (najít citaci). The elevated concentration of growth factors in the area of the lesion will significantly speed up the process of reparation and regeneration - the inflammatory phase is reduced, leukocytes and their cytokines, as well as interleukins are present only in normal, non-elevated concentrations (uvést odkaz). The damaged tissue heals with markedly reduced swelling and the pain is also unambiguously(jednoznačně) reduced which is in virtue of less nociceptive afferentation. The antioedematous effect seems to be the result of an earlier angiogenesis, weak antiendothelial bounds with elevated permeability of proteins and erythrocytes into extracellular space are quickly replaced with adequate endothelial layer, due to the proliferation of endothelium. The healing process is completed with a remodeling of the scar, together with an anticipated reduction of hypertrophic scarring.

ELIGIBILITY:
Inclusion Criteria:

* adult patient (over 18 years old) with deep burn injury indicated for surgery treatment - surgical excisions of devitalised tissue followed by dermoepidermal transplantation
* signed patient´s informed consent

Exclusion Criteria:

* inborn thrombocytopaenia
* haematological malignities
* chronic renal failure (deficiency of platelet´s growth factors)
* not signed patient´s informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-11; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Healing assessed on Vancouver Scar Score | 1st, 3rd, 6th month, 1 and 2 years after surgery
  Vancouver Scar Score is a worldwide measurement tool for assessment of the healing process in the patients with deep burn trauma. It presents us with information regarding the overall healing process.

SECONDARY OUTCOMES:
Percentage of healing | 4th, 6th, 8th, 10th, 12th, 14th, 16th, 18th day after surgery
  The measurements are taken at intervals after the surgical treatment, the calculated data show the percentage of healing compared to the total surgery treatment area (STA) which has been treated with the DE graft and PRP concentrate.
Vitality of the DE graft | 2nd, 4th, 6th, 8th, 10th and 14th post-operative day
  The vitality of the DE graft assessed on a scale enables us to measure the success of the healing process.
Epithelization of the DE graft | 2nd, 4th, 6th, 8th, 10th and 14th post-operative day
  The degree of epithelization assessed on a scale enables us to measure the success of the healing process.
Harvesting surface area | 2nd, 4th, 6th, 8th, 10th and 14th post-operative day
  The state of the harvesting degree area enables us to measure the success of the healing process.

CONTACTS AND LOCATIONS:
Overall Officials: Hana Klosova, MD, Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava-Poruba, Czech Republic, Czechia

REFERENCES:
- [Background] Mehta S, Watson JT. Platelet rich concentrate: basic science and current clinical applications. J Orthop Trauma. 2008 Jul;22(6):432-8. doi: 10.1097/BOT.0b013e31817e793f. PMID 18594311
- [Background] Weibrich G, Kleis WK, Buch R, Hitzler WE, Hafner G. The Harvest Smart PRePTM system versus the Friadent-Schutze platelet-rich plasma kit. Clin Oral Implants Res. 2003 Apr;14(2):233-9. doi: 10.1034/j.1600-0501.2003.140215.x. PMID 12656885
- [Background] Landesberg R, Roy M, Glickman RS. Quantification of growth factor levels using a simplified method of platelet-rich plasma gel preparation. J Oral Maxillofac Surg. 2000 Mar;58(3):297-300; discussion 300-1. doi: 10.1016/s0278-2391(00)90058-2. PMID 10716112
- [Background] Marx RE. Platelet-rich plasma (PRP): what is PRP and what is not PRP? Implant Dent. 2001;10(4):225-8. doi: 10.1097/00008505-200110000-00002. No abstract available. PMID 11813662
- [Background] Mazzucco L, Medici D, Serra M, Panizza R, Rivara G, Orecchia S, Libener R, Cattana E, Levis A, Betta PG, Borzini P. The use of autologous platelet gel to treat difficult-to-heal wounds: a pilot study. Transfusion. 2004 Jul;44(7):1013-8. doi: 10.1111/j.1537-2995.2004.03366.x. PMID 15225241
- [Derived] Prochazka V, Klosova H, Stetinsky J, Gumulec J, Vitkova K, Salounova D, Dvorackova J, Bielnikova H, Klement P, Levakova V, Ocelka T, Pavliska L, Kovanic P, Klement GL. Addition of platelet concentrate to dermo-epidermal skin graft in deep burn trauma reduces scarring and need for revision surgeries. Biomed Pap Med Fac Univ Palacky Olomouc Czech Repub. 2014 Jun;158(2):242-58. doi: 10.5507/bp.2013.070. Epub 2013 Sep 27. PMID 24108222